CLINICAL TRIAL: NCT06983665
Title: Single-Dose, Randomized, Open-Label, Two-Sequence, Two-Period, Double-Crossover, Bioequivalence Study of Liposomal Amphotericin B for Injection in Healthy Chinese Subjects
Brief Title: Human Bioequivalence Study of Liposomal Amphotericin B for Injection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JN-0035-BE01
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Invasive Fungal Infections; Neutropenic Fever; Visceral Leishmaniasis
MeSH Terms: conditions — Invasive Fungal Infections; Febrile Neutropenia; Leishmaniasis, Visceral | interventions — liposomal amphotericin B; Injections; Long-Term Synaptic Depression

STUDY DESIGN:
Masking Description: Open-label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I, Liposomal amphotericin B for injection (Experimental): Test product (Liposomal amphotericin B for injection, Sichuan Huiyu Pharmaceutical Co., Ltd.)
  Interventions: Drug: Test product (Liposomal amphotericin B for injection, Sichuan Huiyu Pharmaceutical Co., Ltd.)
- Group II, AmBisome® (Experimental): Reference product (AmBisome®, Astellas Pharma US Inc.)
  Interventions: Drug: Reference product (AmBisome®, Astellas Pharma US Inc.)

INTERVENTIONS:
Drug: Test product (Liposomal amphotericin B for injection, Sichuan Huiyu Pharmaceutical Co., Ltd.) — Single intravenous administration of 2.0 mg/kg in each period.
  Other Names: Test product.
  Arms: Group I, Liposomal amphotericin B for injection
Drug: Reference product (AmBisome®, Astellas Pharma US Inc.) — Single intravenous administration of 2.0 mg/kg in each period.
  Other Names: Reference product.
  Arms: Group II, AmBisome®

SUMMARY:
A single-center, randomized, open-label, single-dose, two-period, double-crossover study to evaluate the bioequivalence of liposomal amphotericin B for injection (test product) manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd. compared to the reference product (AmBisome®) in healthy Chinese subjects. Secondary objectives include safety evaluation.

DETAILED DESCRIPTION:
The study involves 42 healthy subjects (male and female) aged 18-55 years. Subjects will be randomized into two groups (TR and RT) and receive either the test or reference product in period 1, followed by a 92-day washout period before crossing over to the other product in period 2. Blood samples will be collected at 25 time points for pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participate in the clinical trial, with the ability to sign an informed consent form (ICF) and have a full understanding of trial contents, process, and potential adverse reactions, and be able to understand and adhere to the trial procedures;
2. Chinese male and female subjects aged 18 to 55 years old (inclusive);
3. Male subjects with weight no less than 50.0 kg, and female subjects with weight no less than 45.0 kg. Body mass index (BMI) = weight/height2 (kg/m2). BMI is 18.6-28.5 kg/m2 (both inclusive);
4. At screening, subjects' vital signs, physical examinations, laboratory tests, and electrocardiogram (ECG) results are normal, or abnormal but clinically insignificant as determined by the Investigator;
5. Subjects (including male subjects) have adopted effective contraceptive measures within 14 days prior to the first dosing and are willing to refrain from pregnancy, donating sperm or eggs, and voluntarily use effective contraceptive measures (non-pharmacological contraception during the trial) from the time of signing the informed consent form until 6 months after the last dose.

Exclusion Criteria:

1. Subjects with chronic or severe diseases of the cardiovascular, hepatic, renal, respiratory, hematological and lymphatic, endocrine, immune, mental and nervous, gastrointestinal, metabolic, and skeletal systems, who, as determined by the Investigator, are not suitable to participate in the study;
2. Subjects with clinically significant abnormalities as determined by the Investigator, including physical examination, vital signs, ECG or clinical laboratory tests, especially abnormalities in hepatic and renal functions (subjects with serum creatinine, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) above the upper limit of normal (ULN));
3. Subjects with existing allergic diseases (nettle rash, eczema, etc.), or an atopic constitution (e.g. allergies to two or more medications, foods such as milk, or pollen), or a known history of hypersensitivity to any component of conventional amphotericin B formulations or liposomal amphotericin B formulations, including the active ingredient or any excipients in this product (such as soybean oil), peanuts or soy;
4. Subjects who are positive for any one or more of the following tests: Hepatitis B virus (HBV) surface antigen, hepatitis C virus (HCV) antibody, Treponema pallidum specific antibody and human immunodeficiency virus (HIV) antigen/antibody;
5. Subjects with a history of drug abuse;
6. Subjects who are positive for urine drug screening (methamphetamine (meth), MDMA (ecstasy), THC (cannabis), morphine, ketamine);
7. Regular drinkers within 3 months prior to screening, defined as subjects who drink more than 14 units of alcohol per week (1 unit ≈ 285 mL of beer with 3.5% ABV or 25 mL of spirits with 40% ABV or 85 mL of wine with 10% ABV), or subjects who cannot stop drinking or consuming any alcoholic products throughout the study;
8. Subjects who are positive for breath alcohol test;
9. Subjects with excessive daily consumption of tea, coffee, and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) within the 3 months prior to screening;
10. Subjects with a daily cigarette consumption of > 5 cigarettes/day within 3 months prior to screening, or who cannot discontinue any tobacco-based products, nicotine products, or e-cigarette products throughout the study;
11. Subjects with a history of surgery within 3 months prior to screening, or planned surgery, dental procedures, or hospitalization during the study period;
12. Subjects who have donated blood or experienced massive blood loss (> 400 mL) within 3 months prior to screening, or donated platelets ≥2 therapeutic doses (1 therapeutic dose = 12 U of platelets) within 1 month prior to screening;
13. Subjects who have participated in and received treatment in any drug or medical device clinical study within 3 months prior to screening;
14. Subjects who have received any live vaccine within 3 months prior to screening, or any COVID-19 vaccine within 2 weeks prior to screening, or who are scheduled to be vaccinated within one month after study completion;
15. Subjects who have used any oral contraceptives within 30 days prior to screening or any long-acting estrogen and/or progestin injections and/or implantable contraceptive devices within 6 months prior to screening;
16. Subjects who have used any medications within 28 days prior to screening that affect the absorption and metabolism of the investigational drug (including hepatic enzyme inhibitors, inducers, or those that alter the gastrointestinal environment), or interact with the investigational drug (e.g., corticosteroids, adrenocorticotropic hormone drugs, pyrrolizidine drugs (e.g., ketoconazole, miconazole, clotrimazole, fluconazole), skeletal muscle relaxants, antineoplastic agents, digitalis glycosides, flucytosine, or other nephrotoxic drugs), and who, as determined by the Investigator, are not suitable to participate in the study;
17. Subjects who have used any prescription drugs within 14 days prior to screening or any over-the-counter drugs, Chinese herbal medicines or health products within 7 days prior to screening, except for topical drugs that act on a particular place of body;
18. Subjects who are unable to avoid consuming xanthine-rich beverages (coffee, tea, etc.) or foods (chocolate, animal liver, etc.), or consuming fruits or juices that may affect metabolism (grapefruit, pomelo, mango, dragon fruit, etc.) or iodine-rich foods (seaweed, kelp, etc.) during a period from 48 hours pre-dose to the end of the study, or subjects who have other factors that affect drug absorption, distribution, metabolism and excretion;
19. Subjects who have taken strenuous exercise within 48 hours prior to screening;
20. Subjects who have special requirements for diet and cannot follow the diet provided during the study;
21. Subjects who have difficulty in venous blood collection or a history of fear of needles or hemophobia;
22. Female subjects who are breastfeeding or have a positive pregnancy test result during the screening period or course of the trial;
23. Subjects who, as determined by the Investigator, are not suitable to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax of liposome-encapsulated | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% Cl of Cmax of liposome-encapsulated amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%
Bioequivalence based on AUC0-t of liposome-encapsulated | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% Cl of AUC0-t of liposome-encapsulated amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00% amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%
Bioequivalence based on AUC0-∞ of liposome-encapsulated | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% Cl of AUC0-∞ of liposome-encapsulated amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00% amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00% amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%

SECONDARY OUTCOMES:
Cmax of free amphotericin B | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% Cl of Cmax of free amphotericin B
AUC0-t of free amphotericin B | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% Cl of AUC0-t of free amphotericin B
AUC0-∞ of free amphotericin B | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% Cl of AUC0-∞ of free amphotericin B
Partial exposure indicators (AUC0-10h) of liposome-encapsulated amphotericin B | 0 h before safe dose and 0 h before formal dose to 10 hours post formal dose
  90% Cl of AUC0-10h of liposome-encapsulated amphotericin B
Partial exposure indicators (AUC10-last) of liposome-encapsulated amphotericin B | 10 hours post formal dose to 1320 hours post formal dose
  90% Cl of AUC10-last of liposome-encapsulated amphotericin B
Partial exposure indicators (AUC0-24h) | 0 h before safe dose and 0 h before formal dose to 24 hours post formal dose
  90% Cl of AUC0-24h of free amphotericin B
Partial exposure indicators (AUC24-last) of free amphotericin B | 24 hours post formal dose to 1320 hours post formal dose
  90% Cl of AUC24-last of free amphotericin B
AUC%Extrap | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  Descriptive analysis
Tmax | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  Non-parametric test
t1/2 | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  Descriptive analysis
λz | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  Descriptive analysis
F | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  Descriptive analysis

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, Study Director — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, No.105, Jiefang Road,, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No